CLINICAL TRIAL: NCT05076175
Title: A Phase 2/3, Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Oral Ozanimod (RPC1063) in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis With an Inadequate Response to Conventional Therapy
Brief Title: A Study Investigating Oral Ozanimod (RPC1063) in Pediatric Participants With Moderate to Severe Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM047-001; 2023-509248-86 (Other: EU CTR)
Record Dates: First submitted 2021-10-04; First posted 2021-10-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis; Ozanimod; Pediatric
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ozanimod High Dose (Experimental)
  Interventions: Drug: Ozanimod
- Ozanimod Low Dose (Experimental)
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Other Names: RPC1063

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of ozanimod (RPC1063) in achieving and maintaining clinical remission. Ozanimod will be administered orally to pediatric participants with moderate to severe active ulcerative colitis (UC) who have had an inadequate response to conventional therapy.

ELIGIBILITY:
Inclusion Criteria

* Moderately to severely active Ulcerative Colitis (UC) diagnosed prior to the Screening Visit
* Evidence of UC extending beyond the rectum, as determined by baseline endoscopy
* Has had an inadequate response, loss of response to, or is intolerant to at least 1 of the following treatments for UC: oral aminosalicylates, systemic corticosteroids, immunomodulators, biologic therapy

Exclusion Criteria

* Diagnosis of Crohn's disease or indeterminate colitis
* Has documentation of positive test for toxin producing Clostridium difficile, or polymerase chain reaction examination of the stool
* Apheresis within 2 weeks of randomization
* History of or currently active primary or secondary immunodeficiency, or participants with known genetic disorders as a cause for colitis
* Other protocol-defined inclusion/exclusion criteria apply

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2031-08-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve clinical remission | At Week 52

SECONDARY OUTCOMES:
Proportion of participants who achieve clinical remission | At Week 10
Proportion of participants who achieve clinical response | At Week 52
Proportion of participants who achieve clinical response | At Week 10
Proportion of participants who achieve symptomatic remission | At Week 10 and Week 52
Time to achievement of symptomatic remission | Up to 6 years
Proportion of participants who achieve endoscopic improvement | At Week 10 and Week 52
Proportion of participants who achieve corticosteroid free remission | At Week 52
Incidence of Adverse Events (AEs) | Up to 6 years
Incidence of Serious Adverse Events | Up to 6 years
Incidence of AEs leading to discontinuation from treatment | Up to 6 years
Incidence of AEs of special interest (AESIs) | Up to 6 years
Steady state systemic exposure of ozanimod and CC112273 | At Week 18 and throughout the study, up to 70 weeks
Absolute change from baseline in Absolute Lymphocyte Count (ALC) | Up to 6 years
Percent change from baseline in ALC | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (36):
  - Local Institution - 0041, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Local Institution - 0052, Garden Grove, California
  - Loma Linda University Health System, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Local Institution - 0096, Sacramento, California
  - Local Institution - 0007, Hartford, Connecticut
  - Local Institution - 0064, Washington D.C., District of Columbia
  - Local Institution - 0075, Orlando, Florida
  - Local Institution - 0016, Atlanta, Georgia
  - Local Institution - 0101, Park Ridge, Illinois
  - Local Institution - 0100, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Partners, Portland, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - Local Institution - 0042, Springfield, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Local Institution - 0028, New York, New York
  - Columbia University Medical Center, New York, New York
  - Local Institution - 0023, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Local Institution - 0047, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution - 0062, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Local Institution - 0099, Charleston, South Carolina
  - Local Institution - 0103, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Local Institution - 0091, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Local Institution - 0086, Murdoch, Western Australia
- Belgium (6):
  - Local Institution - 0076, Brussels, Bruxelles-Capitale, Région de
  - UZ Leuven, Leuven, Vlaams-Brabant
  - UZ Brussel, Brussels
  - Local Institution - 0063, Edegem
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Local Institution - 0071, Liège
- Canada (3):
  - Local Institution - 0083, Hamilton, Ontario
  - Local Institution - 0104, Toronto, Ontario
  - Local Institution - 0082, Toronto, Ontario
- France (5):
  - CHU de Toulouse - Hôpital des Enfants, Toulouse, Haute-Garonne
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre, Caen
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Local Institution - 0073, Paris
- Germany (3):
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
- Israel (3):
  - Schneider Children's Medical Center, Petah Tikva, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
- Japan (10):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Komatsu Municipal Hospital, Komatsu, Ishikawa-ken
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Institute of Science Tokyo Hospital, Bunkyo-Ku, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Juntendo University Hospital, Tokyo
- Poland (9):
  - Local Institution - 0084, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
  - Centrum Zdrowia Dziecka w Warszawie, Warsaw, Masovian Voivodeship
  - Local Institution - 0015, Rzeszów, Podkarpackie Voivodeship
  - Local Institution - 0013, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0079, Gdansk, Pomeranian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - Local Institution - 0092, Lodz, Łódź Voivodeship
- Local Institution - 0098, San Juan, Puerto Rico
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Moskva
- Spain (5):
  - Local Institution - 0048, Badalona, Barcelona [Barcelona]
  - Local Institution - 0051, Esplugues de Llobregat, Barcelona [Barcelona]
  - Local Institution - 0044, Madrid, Madrid, Comunidad de
  - Local Institution - 0057, Madrid
  - Local Institution - 0050, Madrid
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham, England
  - King's College Hospital, London, Greater London
  - Barts Health NHS Trust, London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05076175.html